CLINICAL TRIAL: NCT03178045
Title: Ambulatory Cancer Care Electronic Symptom Self-Reporting for Surgical Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Brigham and Women's Hospital (Other); University of Rochester (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 17-293
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Results first posted 2020-11-17 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Patient Reported Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Team Monitoring: Team Monitoring is the current standard of care for patients at Josie Robertson Surgery Center (JRSC).
  Interventions: Other: Team Monitoring
- Enhanced Feedback: The electronic system will provide tailored normative data visualizations that offer context and education to patients regarding expected symptom severity.
  Interventions: Other: Enhanced Feedback

INTERVENTIONS:
Other: Team Monitoring — In this cohort, the electronic system will provide advanced informatics support for push notifications to the care team based on the severity of the symptoms reported. This platform promotes early detection and intervention. The care team is alerted when patients experience symptoms out of the expected range or if symptoms are worsening. Nurses receive secure message notifications and will contact the patient by phone depending on symptom severity. If a patient responds with a moderate-severe answer, the office team gets an alert and calls the patient during business hours.
  Groups: Team Monitoring
Other: Enhanced Feedback — In this cohort, the electronic system will provide tailored normative data visualizations that offer context and education to patients regarding expected symptom severity. The information provided to patients in the Enhanced Feedback group will be procedure specific and based on continuously updated PRO-CTCAE data from previous patients. Patients are thus able to see their own recovery trajectory relative to that of patients who have undergone the same procedure. Care is patient activated in that patients will use the information about expected symptoms to decide whether they should call the care team (e.g., if they are experiencing symptoms that are more severe or more prolonged than expected). If a patient reports severe symptoms, they are instructed to immediately contact their physician's office or seek medical attention.
  Groups: Enhanced Feedback

SUMMARY:
The aim of this study is to understand and improve the experience of patients after surgery by comparing two methods of following symptoms while the patient recovers at home.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years of age who are scheduled for ambulatory cancer surgery at JRSC and their caregivers will be eligible for study participation.

Exclusion Criteria:

* Inability to speak English
* Inability to access a computer, tablet, or mobile phone
* For patients: not interested in/unable to sign up for the MyMSK Patient Portal
* For caregivers: Unable to provide an email address
* Cognitive impairment that prohibits informed consent or understanding of the study protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who are scheduled for surgery at Josie Robertson Surgery Center (JRSC).
Sampling Method: Probability Sample
Enrollment: 2793 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Allen, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stabile C, Temple LK, Ancker JS, Basch E, Carter J, Miranda M, Stein D, Stetson PD, Vickers A, Simon BA, Pusic AL. Ambulatory cancer care electronic symptom self-reporting (ACCESS) for surgical patients: a randomised controlled trial protocol. BMJ Open. 2019 Sep 17;9(9):e030863. doi: 10.1136/bmjopen-2019-030863. PMID 31530612
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Team Monitoring: Team monitoring is the current standard of care for patients at the Josie Robertson Surgical Center (JRSC) at Memorial Sloan Kettering Cancer Center (MSK). Patients report their symptoms via an electronic questionnaire called the Recovery Tracker, delivered through an in-house informatics platform known as the ambulatory cancer care electronic symptom self-reporting (ACCESS) system. The healthcare team receives portal-secure message alerts if patients report symptoms above a specified threshold and contact the patient by phone during business hours. Given the need for real-time feedback for some symptoms, patients who report very severe symptoms receive a bold red alert instructing them to immediately contact their care team or seek medical attention.
- Enhanced Feedback: In the enhanced feedback cohort, the ACCESS system provides tailored normative data visualizations that offer context and education to patients regarding expected symptom severity. The feedback report consists of periodically updated PRO data from previous patients that are stratified by surgical procedure and postoperative date. As a result, patients can see their recovery trajectories relative to others who have undergone the same procedure. Care is 'patient-activated', in that patients use the information about expected symptoms to decide whether they should call the care team, for instance, if they experience symptoms that are more severe or more prolonged than expected. Similar to the team monitoring cohort, patients who report very severe symptoms are instructed to immediately contact their physician's office, and the care team receives an alert.
Period: Overall Study
Arm/Group | Team Monitoring | Enhanced Feedback
Started | 1396 | 1397
Completed | 1310 | 1314
Not Completed | 86 | 83
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Surgery Cancelled/Relocated | 34 | 30
Not completed — Procedure Ineligible Post-Operatively/Pr | 47 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Team Monitoring | Enhanced Feedback | Total
Number analyzed (Participants) | 1,310 | 1,314 | 2624
Age, Continuous [Median (Full Range); unit: years] | 54 [20 to 86] | 54 [22 to 83] | 54 [20 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 948 | 933 | 1881
  Male | 362 | 381 | 743
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 80 | 86 | 166
  Not Hispanic or Latino | 1146 | 1163 | 2309
  Unknown or Not Reported | 84 | 65 | 149
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 80 | 78 | 158
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 74 | 96 | 170
  White | 1073 | 1045 | 2118
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 81 | 91 | 172
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1310 | 1314 | 2624

OUTCOME MEASURES:

1. Primary Outcome: Rates of UCC Visits and Readmissions Between the Team Monitoring and Enhanced Feedback Cohorts up to 30 Days Post-operatively
Description: To compare the effectiveness of Team Monitoring and Enhanced Feedback with regard to urgent care, emergency department visits, and readmissions up to 30 days post-operatively.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Team Monitoring | Enhanced Feedback
Number analyzed (Participants) | 1,310 | 1,314
Participants
  UCC with Readmission within 30 days | 31 | 38
  UCC without Readmission within 30 days | 44 | 60
  Readmission within 30 days | 32 | 39
  No UCC or Readmissions within 30 days | 1203 | 1177

2. Secondary Outcome: Difference in Total Number of Nursing Follow-up Calls Between Team Monitoring and Enhanced Feedback Cohorts up to 30 Days Post-Operatively
Description: To evaluate the difference in nursing phone calls between each study arm up to 30 days post-operatively.
Time Frame: 30 days post-operatively
Measure: Mean (Standard Deviation); unit: Nursing Calls
Arm/Group | Team Monitoring | Enhanced Feedback
Number analyzed (Participants) | 1310 | 1314
Nursing Calls | 3.79 (3.14) | 3.40 (2.71)

3. Secondary Outcome: Differences in Total Number of Unplanned Clinic Visits Between Team Monitoring and Enhanced Feedback Cohorts Up to 30 Days Post-Operatively
Description: To evaluate the difference in unplanned clinic visits and phone referrals to clinic between each study arm up to 30 days post-operatively.
Time Frame: 30 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Team Monitoring | Enhanced Feedback
Number analyzed (Participants) | 1310 | 1314
Participants
  0 Clinic Visits | 349 | 347
  1 Clinic Visit | 467 | 476
  2 Clinic Visits | 301 | 282
  3 Clinic Visits | 129 | 137
  4 Clinic Visits | 49 | 52
  5 Clinic Visits | 9 | 15
  6 Clinic Visits | 5 | 4
  7 Clinic Visits | 0 | 1
  8 Clinic Visits | 1 | 0
Statistical Analysis 1: Comparison: Team Monitoring; Test type: Other — Multivariable Logistic Regression; Estimated Increase = 0.23, 95% CI 2-sided [-3.1 to 3.6]

4. Secondary Outcome: Differences in Total Number of Pain Management Referrals Between Team Monitoring and Enhanced Feedback Cohorts Up to 30 Days Post-Operatively
Description: To evaluate the difference in pain management referrals between each study arm up to 30 days post-operatively.
Time Frame: 30 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Team Monitoring | Enhanced Feedback
Number analyzed (Participants) | 1310 | 1314
Participants
  0 Clinic Visit | 1299 | 1302
  1 Clinic Visit | 10 | 11
  2 Clinic Visits | 1 | 1
Statistical Analysis 1: Comparison: Team Monitoring; Test type: Other — Multivariable logistic regression; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.69 to 1.31]

5. Secondary Outcome: Differences in Adverse Events Between Team Monitoring and Enhanced Feedback Cohorts Up to 30 Days Post-Operatively
Description: To evaluate the difference in adverse events between each study arm up to 30 days post-operatively.
Time Frame: 30 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Team Monitoring | Enhanced Feedback
Number analyzed (Participants) | 1310 | 1314
Participants
  0 Adverse Events | 1260 | 1258
  1 Adverse Event | 47 | 56
  2 Adverse Events | 3 | 0
Statistical Analysis 1: Comparison: Team Monitoring; Test type: Other — Longitudinal mixed effects regression; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.60 to 1.32]

6. Secondary Outcome: Interaction in Participants Anxiety Measured by 3 Items on the Patient Reported Outcome Common Terminology Criteria for Adverse Events Survey (PRO-CTCAE)
Description: This analysis utilized 3 anxiety items from the PRO-CTCAE survey. The responses were defined on a scale of 0-4 with higher scores representing stronger agreement with the item (higher anxiety). The 3 items were summed to generate an overall score ranging from 0-12. 139 patients responded to only some of the 3 items and were counted as a missing value for the overall sum score. As the surveys were repeated daily, longitudinal mixed effects regression was used to test the association between the anxiety sum score and randomization arm after adjusting for time, randomization strata, and an interaction between randomization arm and time with a random intercept for patient.
Time Frame: 10 days post-operatively
Measure: Mean (95% Confidence Interval); unit: reduction in anxiety score
Groups:
- Difference in Participants Anxiety: Difference in Participants Anxiety Measured by PROCTCAE Survey
Arm/Group | Team Monitoring | Enhanced Feedback | Difference in Participants Anxiety
Number analyzed (Participants) | 1310 | 1314 | 2624
reduction in anxiety score
  Post-Op Day 2 | 0.03 [0.02 to 0.05] | 3.0 [2.8 to 3.3] | 0.15 [-0.07 to 0.35]
  Post-Op Day 3 | 2.9 [2.7 to 3.1] | 2.9 [2.7 to 3.1] | 0.11 [-0.09 to 0.31]
  Post-Op Day 4 | 2.8 [2.6 to 3.0] | 2.8 [2.6 to 3.0] | 0.07 [-0.12 to 0.26]
  Post-Op Day 5 | 2.7 [2.5 to 2.9] | 2.7 [2.5 to 2.9] | 0.03 [-0.15 to 0.21]
  Post-Op Day 6 | 2.6 [2.4 to 2.8] | 2.6 [2.4 to 2.8] | -0.01 [-0.18 to 0.16]
  Post-Op Day 7 | 2.5 [2.3 to 2.7] | 2.5 [2.3 to 2.7] | -0.05 [-0.22 to 0.12]
  Post-Op Day 8 | 2.5 [2.3 to 2.7] | 2.4 [2.2 to 2.6] | -0.08 [-0.26 to 0.08]
  Post-Op Day 9 | 2.4 [2.2 to 2.6] | 2.3 [2.1 to 2.5] | -0.12 [-0.30 to 0.04]
  Post-Op Day 10 | 2.3 [2.1 to 2.5] | 2.2 [1.9 to 2.4] | -0.16 [-0.35 to 0.01]

7. Secondary Outcome: Differences in Patient Engagement Between Cohorts at 14 Days Post-Operatively Utilizing the Patient Activation Measure (PAM) and Adjusting for Strata and Pre-Operative PAM Score
Description: To evaluate the difference in patient engagement between each study arm at 14 days post-operatively adjusting for strata and preoperative PAM overall score. The survey consists of 10 items with five response options: strongly disagree, disagree, undecided, agree and strongly agree defined on a scale of 1-5 with higher scores representing stronger agreement with the item. The items in the PAM survey were combined to generate an overall mean score at each timepoint - a theoretical score of 0-100. A higher score indicates stronger patient engagement. If a patient is missing a response to an item(s), the overall score is considered missing for that patient/timepoint. Participants who answered the survey were included in this analysis. 560 patients were analyzed in the Team Monitoring Arm and 541 were analyzed in the Enhanced Feedback Arm.
Time Frame: 14 days post-operatively
Measure: Mean (Standard Deviation); unit: PAM Score at 14 Days
Arm/Group | Team Monitoring | Enhanced Feedback
Number analyzed (Participants) | 560 | 541
PAM Score at 14 Days | 3.39 (0.40) | 3.37 (0.43)

8. Secondary Outcome: Differences in Patient Engagement Between Team Monitoring and Enhanced Feedback Cohorts at 60 Days Post-Operatively Utilizing the Patient Activation Measure (PAM) and Adjusting for Strata and Pre-Operative PAM Score
Description: To evaluate the difference in patient engagement between each study arm 60 days post-operatively adjusting for strata and preoperative PAM overall score. The survey consists of 10 items with five response options: strongly disagree, disagree, undecided, agree and strongly agree defined on a scale of 1-5 with higher scores representing stronger agreement with the item. The items in the PAM survey were combined to generate an overall mean score at each timepoint - a theoretical score of 0-100. A higher score indicates stronger patient engagement. If a patient is missing a response to an item(s), the overall score is considered missing for that patient/timepoint. 465 participants form the Team Monitoring Arm and 460 participants from the Enhanced Feedback arm were analyzed who answered the Patient Activation Measure at POD 60.
Time Frame: 60 days post-operatively
Measure: Mean (Standard Deviation); unit: PAM Score at 60 Days
Arm/Group | Team Monitoring | Enhanced Feedback
Number analyzed (Participants) | 465 | 460
PAM Score at 60 Days | 3.47 (0.40) | 3.44 (0.44)

9. Secondary Outcome: Differences in Caregiver Burden Between Team Monitoring and Enhanced Feedback Cohorts Utilizing the Caregiver Reaction Assessment (CRA).
Description: To evaluate the difference in caregiver burden between each study arm at two timepoints: 14 days post-operatively. Scoring information for the CRA: The Caregiver Reaction Assessment involved 24 items given at 14 days and repeated at 60 days with the following potential responses: strongly disagree, disagree, undecided, agree, and strongly agree which we defined on a scale of 1-5 with higher scores representing stronger agreement with the item. These items are combined into 5 subscales: health problems, financial problems, lack of family support, disrupted schedule, and self-esteem. For each subscale, a total score was computed as the average of the subsequent item scores, with a range between 1 and 5. A higher score represented a stronger agreement with the attribute.
Time Frame: 14 days post-operatively
Measure: Mean (Standard Deviation); unit: score on CRA
Arm/Group | Team Monitoring | Enhanced Feedback
Number analyzed (Participants) | 1310 | 1314
score on CRA
  Health Problems | 2.40 (0.46) | 2.45 (0.52)
  Financial Problems | 1.76 (0.85) | 1.78 (0.88)
  Lack of Family Support | 1.59 (0.61) | 1.75 (0.66)
  Disrupted Schedule | 2.72 (0.88) | 2.70 (0.86)
  Self Esteem | 4.52 (0.35) | 4.47 (0.35)

10. Secondary Outcome: Differences in Caregiver Burden Between Team Monitoring and Enhanced Feedback Cohorts Utilizing the Caregiver Reaction Assessment (CRA).
Description: To evaluate the difference in caregiver burden between each study arm at two timepoints: 60 days post-operatively. Scoring information for the CRA: The Caregiver Reaction Assessment involved 24 items given at 14 days and repeated at 60 days with the following potential responses: strongly disagree, disagree, undecided, agree, and strongly agree which we defined on a scale of 1-5 with higher scores representing stronger agreement with the item. These items are combined into 5 subscales: health problems, financial problems, lack of family support, disrupted schedule, and self-esteem. For each subscale, a total score was computed as the average of the subsequent item scores, with a range between 1 and 5. A higher score represented a stronger agreement with the attribute.
Time Frame: 60 days post-operatively
Measure: Mean (Standard Deviation); unit: score on CRA
Arm/Group | Team Monitoring | Enhanced Feedback
Number analyzed (Participants) | 1310 | 1314
score on CRA
  Health Problems | 2.34 (0.47) | 2.44 (0.50)
  Financial Problems | 1.93 (0.91) | 1.90 (0.90)
  Lack of Family Support | 1.71 (0.65) | 1.76 (0.73)
  Disrupted Schedule | 2.43 (0.93) | 2.43 (0.87)
  Self Esteem | 4.45 (0.36) | 4.42 (0.41)

ADVERSE EVENTS:
Time Frame: 30 days post-operative
Arm/Group | Team Monitoring | Enhanced Feedback
All-Cause Mortality (participants affected / at risk) | 0/1310 | 0/1314
Serious Adverse Events (participants affected / at risk) | 0/1310 | 0/1314
Other Adverse Events (participants affected / at risk) | 0/1310 | 0/1314

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT03178045/Prot_SAP_000.pdf